CLINICAL TRIAL: NCT03603470
Title: Total Hip Arthroplasty Instability and Lumbo-pelvic Kinematics: EOS Imaging Assessment of Variation in Spinal and Pelvic Parameters From Standing to Sitting
Acronym: HIPEOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AOIGCSMERRI/2017/PK-01
Record Dates: First submitted 2018-07-02; First posted 2018-07-27 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with previous prothesis instability (Other)
  Interventions: Other: EOS imagery
- Patients without prothesis instability (Other)
  Interventions: Other: EOS imagery

INTERVENTIONS:
Other: EOS imagery — Whole body EOS imaging in seated and standing position

SUMMARY:
The authors hypothesize that a pelvic kinematic disorder, demonstrated by a significant decrease in sacral slope, is associated with the risk of instability of total hip prosthesis, the sacral slope being measured by an EOS imaging system during the transition to sitting in unstable patients versus patients with no history of instability.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient must be at least 18 years old and less than 85 years old
* Patient has a conventional first intention total hip arthroplasty (not dual mobility) by posterior approach
* "Case" patients have at least one previous episode of prosthetic dislocation repaired with surgery
* "Control" patients have no previous episode of prosthetic dislocation with more than 2 year since initial intervention

Exclusion Criteria:

* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient is pregnant, parturient or breastfeeding
* Patient with lumbar instrumentation
* Patient with severe dementia (Mini Mental State Examination < 10)
* Patient with American Society of Anesthesiologists score ≥ 4
* Patient experience multiple falls
* Patient requiring early revision surgery (<15 days postoperatively
* Patient with obvious implant positioning error on an X-ray of the pelvis.
* Patient with dislocation of traumatic origin (significant kinetic trauma)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Sacral slope between standing to sitting difference between groups | Day 0
  Sacral slope between standing to sitting difference between groups
Rate of type 1 pelvic kinematic disorder between groups | Day 0
  Measured by sacral slope difference from standing to seated position < 12°.

SECONDARY OUTCOMES:
Lumbar lordosis between standing and seating between groups | Day 0
  degree
Femoroacetabular flexion between standing and seating between groups | Day 0
  degree
Lewinnek plane (Anterior pelvic plane) between standing and seating between groups | Day 0
  degree
Pelvic version between standing and seating between groups | Day 0
  degree
Classification of patients' pelvic kinematic disorder (Type 1 or 2) | Day 0
  Type 1 = Difference in sacral slope between standing and seated position < 12° Type 2 = pelvic version < 20° standing
Classification of patients according to pelvic incidence | Day 0
  Presence/absence
Classification of patients according to sacral slope | Day 0
  Presence/absence
Classification of patients according to sagittal imbalance | Day 0
  Presence/absence of: Sagittal Vertical Axis > 50 mm; Spino-Sacral Angle < 127°
Evolution of acetabular positioning (anteversion and inclination in degree) from standing to sitting | Day 0
  Degree

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Kouyoumdjian, MD, Principal Investigator — CHU Nimes
Locations (2):
- France (2):
  - CHU Lapeyronie de Montpellier, Montpellier
  - CHU Nimes, Nîmes